CLINICAL TRIAL: NCT01293617
Title: Blackberry Intake and Biomarkers of Cancer Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Janet A. Novotny, Ph.D., Beltsville Human Nutrition Research Center, USDA
Organization: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS36
Record Dates: First submitted 2011-01-24; First posted 2011-02-10 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Gelatin

ARMS (2):
- Gelatin (Placebo Comparator)
  Interventions: Other: Gelatin
- Blackberries (Experimental)
  Interventions: Other: Blackberries

INTERVENTIONS:
Other: Blackberries — 300 g blackberries daily for 5 days
  Arms: Blackberries
Other: Gelatin — 300 g gelatin per day for 5 days
  Arms: Gelatin

SUMMARY:
Berry components have been shown to influence cancer processes in cell culture studies. The investigators will conduct a study to investigate if blackberries influence the same cancer processes in a human feeding study.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking men and women
* Aged 40-75
* BMI 19-38 kg/m2

Exclusion Criteria:

* Younger then 40 ears old or older than 75 years old
* BMI less than 19 or greater than 38
* Use of blood-thinning medications such as warfarin, dicumarol, or anisinidione
* Presence of kidney disease, liver disease, gout, certain cancers, untreated thyroid, gastrointestinal, other metabolic diseases or malabsorption syndromes
* Type 2 diabetes requiring the use of oral antidiabetic agents or insulin
* Fasting triglycerides greater than 300 mg/dL
* Fasting glucose greater than 126 mg/dL
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g. vegetarians, very low fat diets, high protein diets)
* Use of prescription of over-the-counter antiobesity medications or supplements during and for at least 6 months prior to the start of the study or a history of a surgical intervention for obesity
* Active cardiovascular disease
* Use of any tobacco products in the past 6 months
* Use of oral or IV antibiotics during the month preceding the study or during the study
* Unwillingness to abstain from vitamin, mineral, and herbal supplements for two weeks prior to the start of the study
* Known (self-reported) allergy or adverse reaction to blackberries or gelatin
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 8-oxo-dG levels after 5 days | Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Janet A Novotny, Ph.D., Principal Investigator — Beltsville Human Nutrition Research Center, USDA
Locations (1):
- Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

REFERENCES:
- See also: Recruiting Info — http://ars.usda.gov/Research/docs.htm?docid=18347&page=2